CLINICAL TRIAL: NCT01729468
Title: Prevention of Pre-eclampsia and SGA by Low-Dose Aspirin in Nulliparous Women With Abnormal First-trimester Uterine Artery Dopplers
Acronym: PERASTUN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PHRN08-FP/PERASTUN; 2011-003536-30 (EudraCT Number); 2012-R8 (Other: CPP); A120316-72 (Other: Afssaps); 912140 (Other: CNIL)
Record Dates: First submitted 2012-11-02; First posted 2012-11-20 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Pre-eclampsia; Intra-uterine Growth Restriction
Keywords: Low Dose Acetylsalicylic Acid; Prevention; Pre-eclampsia; Intra-uterine Growth Restriction; Primiparous Women; Bilateral Uterine Artery Notches; First Quarter
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Experimental): Aspirin 160 mg per day
  Interventions: Drug: Aspirin
- Placebo (Placebo Comparator): Placebo 160 mg per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — Aspirin, 160 mg per day until 34 weeks of gestation
  Arms: Aspirin
Drug: Placebo — Placebo, 160 mg per day until 34 weeks of gestation
  Arms: Placebo

SUMMARY:
The objective of this study is to test the efficacy of low-dose aspirin (160 mg/day), given bedtime and started early during pregnancy (≤ 15 +6 weeks of gestation) in nulliparous pregnant women selected as "high-risk" by the presence of a bilateral uterine artery notch and/or bilateral uterine artery PI ≥ 1.7 during the first trimester ultrasound scan (11-13+6 weeks), to prevent the occurrence of pre-eclampsia or small for gestational age at birth.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Nulliparous (no previous pregnancy ≥ 22 SA)
* Singleton pregnancy
* Gestational age ≤ 15 +6 weeks
* Bilateral uterine artery notch (grade ≥ 2) and/or bilateral uterine artery PI ≥ 1.7 during first trimester ultrasound (CRL between 45 and 84 mm)
* Maternal informed consent obtained
* Affiliated to social security system

Exclusion Criteria:

* Women considering voluntary pregnancy termination (≤ 14 weeks)
* Pre-existing (maternal) indication for premature delivery before 37 weeks
* Fetal condition detected during the first trimester scan (fetal malformation or nuchal translucency ≥ 95th percentile)
* Women under anticoagulation
* Allergy or hypersensitivity to Kardegic® or one of its constituents
* Secondary hemostasis disorder responsible for bleeding or risk of bleeding
* Peptic ulcer under evolution
* Lupus or antiphospholipid syndrome

Min Age: 18 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1106 (Actual)
Dates: Start 2012-06-27 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2016-10-25 (Actual)

PRIMARY OUTCOMES:
Preeclampsia (diagnosed per ACOG criteria) and small for gestational age at birth (≤5th percentile on customized growth curves) | women will be followed for the duration of pregnancy and postpartum, an expected average of 26 to 31 weeks

SECONDARY OUTCOMES:
Small for gestational age at birth (≤5th percentile on customized growth curves) | women will be followed for the duration of pregnancy, an expected average of 25 to 30 weeks
Pre-eclampsia (ACOG criteria) requiring delivery before 34 weeks | women will be followed for the duration of pregnancy and postpartum, an expected average of 26 to 31 weeks
Severe pre-eclampsia (ACOG criteria) | women will be followed for the duration of pregnancy and postpartum, an expected average of 26 to 31 weeks
Perinatal death (22 weeks of gestation to 7 days postnatal) | women will be followed for the duration of pregnancy and postpartum, an expected average of 26 to 31 weeks
Pre-eclampsia (ACOG criteria) | women will be followed for the duration of pregnancy and postpartum, an expected average of 26 to 31 weeks
Adverse effects of treatment | women will be followed for the duration of pregnancy and postpartum, an expected average of 26 to 31 weeks

OTHER OUTCOMES:
Mode of delivery (vaginal or cesarean) | women will be followed for the duration of pregnancy, an expected average of 25 to 30 weeks
Mode of anesthesia for delivery | women will be followed for the duration of pregnancy, an expected average of 25 to 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Franck PERROTIN, MD-PhD, Principal Investigator — University Hospital, Tours
Locations (17):
- France (16):
  - Service de Gynécologie-Obstétrique, Groupe Hospitalier Pellegrin, CHRU de Bordeaux, Bordeaux
  - Service de Gynécologie-Obstétrique, HFME, Hospices Civils de Lyon, Bron
  - Service de gynécologie-obstétrique, Polyclinique du PARC, Caen
  - Service de Gynécologie-Obstétrique, Hôpital d'Estaing, CHU de Clermont-Ferrand, Clermont-Ferrand
  - Service de gynécologie-obstétrique, Hôpital Couple Enfant, CHRU de Grenoble, Grenoble
  - Cabinet Mosaïque Santé, La Chaussée-Saint-Victor
  - Service de gynécologie-obstétrique, CHR Le Mans, Le Mans
  - Service de Gyénécologie-Obstétrique, Hôpital Jeanne de Flandre, CHRU de Lille, Lille
  - Service de Gynécologie-Obstétrique, Hôpital Arnaud de Villeneuve, CHRU de Montpellier, Montpellier
  - Service de gynécologie-obstétrique, Hôpital Mère-Enfant, CHRU de Nantes, Nantes
  - Service de gynécologie-obstétrique, Polyclinique de l'Atlantique, Nantes
  - Service de Gynécologie-Obstétrique, Hôpital Carémeau, CHRU de Nîmes, Nîmes
  - Service de Gynécologie-Obstétrique, Hôpital Porte Madeleine, CHR d'Orléans, Orléans
  - Centre de dépistage PRIMA FACIE, Hôpital Necker, APHP, Paris
  - Service de Gynécologie-Obstétrique, Hôpital Paule de Viguier, CHU de Toulouse, Toulouse
  - Service de Gynécologie-Obstetrique, Centre Olympe de Gouges, CHRU de Tours, Tours
- Service de gynécologie-obstétrique, Maison de la Femme de la Mère et de l'Enfant, CHU de Fort de France, Fort-de-France, Martinique

REFERENCES:
- [Background] Poon LC, Syngelaki A, Akolekar R, Lai J, Nicolaides KH. Combined screening for preeclampsia and small for gestational age at 11-13 weeks. Fetal Diagn Ther. 2013;33(1):16-27. doi: 10.1159/000341712. Epub 2012 Sep 13. PMID 22986844
- [Background] Ayala DE, Ucieda R, Hermida RC. Chronotherapy with low-dose aspirin for prevention of complications in pregnancy. Chronobiol Int. 2013 Mar;30(1-2):260-79. doi: 10.3109/07420528.2012.717455. Epub 2012 Sep 24. PMID 23004922
- [Background] Plasencia W, Maiz N, Poon L, Yu C, Nicolaides KH. Uterine artery Doppler at 11 + 0 to 13 + 6 weeks and 21 + 0 to 24 + 6 weeks in the prediction of pre-eclampsia. Ultrasound Obstet Gynecol. 2008 Aug;32(2):138-46. doi: 10.1002/uog.5402. PMID 18634131
- [Result] Diguisto C, Le Gouge A, Marchand MS, Megier P, Ville Y, Haddad G, Winer N, Arthuis C, Doret M, Debarge VH, Flandrin A, Delmas HL, Gallot D, Mares P, Vayssiere C, Sentilhes L, Cheve MT, Paumier A, Durin L, Schaub B, Equy V, Giraudeau B, Perrotin F; Groupe de Recherche en Obstetrique et Gynecologie (GROG). Low-dose aspirin to prevent preeclampsia and growth restriction in nulliparous women identified by uterine artery Doppler as at high risk of preeclampsia: A double blinded randomized placebo-controlled trial. PLoS One. 2022 Oct 19;17(10):e0275129. doi: 10.1371/journal.pone.0275129. eCollection 2022. PMID 36260615